CLINICAL TRIAL: NCT01400048
Title: Aloe Vera Versus Placebo for Patients With Irritable Bowel Syndrome
Brief Title: Aloe Vera in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Calmino group AB (Unknown)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aloe Vera AVH200
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aloe vera effervescent tablet (AVH200) (Active Comparator)
  Interventions: Dietary Supplement: Aloe vera effervescent tablet (AVH200)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Aloe vera effervescent tablet (AVH200) — 250 mg aloe vera and 60 mg ascorbic acid, Aloe Life®
  Arms: Aloe vera effervescent tablet (AVH200)
Dietary Supplement: Placebo control — 60mg Ascorbic acid
  Arms: Placebo

SUMMARY:
The purpose of the present study is to study the effect of aloe vera in the treatment of IBS patients in a randomized, double-blind placebo controlled study.

DETAILED DESCRIPTION:
There is limited knowledge of the IBS pathophysiology, absence of biological markers and therefore few effective treatment options. IBS therefore contributes to difficulties in the management of the patients. Aloe vera has a long association with herbal medicine, from the Ebers Papyrus from 16th century BCE. It is alleged to be effective in treatment of wounds, to improve blood glucose levels in diabetics, and it may reduce symptoms and inflammation in patients with ulcerative colitis. Evidence of the effects of aloe vera in the treatment of IBS, is however limited and contradictory.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to the Rome III criteria
* Adults

Exclusion Criteria:

* other GI disorders
* other medical conditions
* were pregnancy or breast-feeding
* food allergy or intolerance to other than lactose
* ongoing intake of aloe vera products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
IBS symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, MD, PhD, Principal Investigator — Dept of Internal medicine, Sahlgrenska UH, Gothenburg, Sweden
Locations (1):
- Mag-tarmlab, Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Ahluwalia B, Magnusson MK, Bohn L, Storsrud S, Larsson F, Savolainen O, Ross A, Simren M, Ohman L. Randomized clinical trial: Effects of Aloe barbadensis Mill. extract on symptoms, fecal microbiota and fecal metabolite profiles in patients with irritable bowel syndrome. Neurogastroenterol Motil. 2020 Aug;32(8):e13860. doi: 10.1111/nmo.13860. Epub 2020 Apr 20. PMID 32314514